CLINICAL TRIAL: NCT01792336
Title: Gamma Frequency Transcranial Magnetic Stimulation in Dystonia
Brief Title: Transcranial Magnetic Stimulation for Focal Hand Dystonia
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130076; 13-N-0076
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-02-19

CONDITIONS: Dystonia
Keywords: Repetitive TMS (rTMS); Transcranial Magnetic Stimulation (TMS); Motor Cortex; Focal Hand Dystonia; Facilitation
MeSH Terms: conditions — Dystonia; Dystonia, Focal, Task-Specific

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* The brain has natural electrical rhythms of brain activities. These rhythms may be different in people with movement disorders, such as dystonia (involuntary muscle movement, cramps, or tremors). Understanding these rhythms may provide more information about movement disorders.
* Focal hand dystonia, also known as "writer's cramp" or "musician's cramp," is a painful condition that affects the hand and arm muscles. Researchers want to use transcranial magnetic stimulation (TMS) to study brain rhythms in people with and without focal hand dystonia.

Objectives:

- To better understand brain rhythms involved in focal hand dystonia.

Eligibility:

* Individuals between 18 and 70 years of age who are right-handed and have focal hand dystonia.
* Healthy right-handed volunteers between 18 and 60 years of age.

Design:

* Participants will be screened with a physical exam and medical history.
* This study includes two tests: a pilot test and a main test. The pilot test will determine the frequency of TMS that will be used in the main test. Participants may be in one or both tests. Each test requires a single outpatient visit that will last up to 5 hours.
* Participants will have a base test to see how their muscles respond to TMS. This will look at the electrical activity of the muscles. Participants will have a wire coil held on their scalp. A brief electrical current will pass through the coil. It creates a magnetic pulse that stimulates the brain. Researchers will test the TMS on the right and left sides of the head. This will help find the spot that activates the finger muscles, and see how much TMS is needed.
* In the main test, participants will have repetitive TMS (rTMS). rTMS involves repeated magnetic pulses delivered in short bursts. There will be four pulses in each burst. Participants will have multiple bursts during the test. This test will look at how the muscles of the hand and fingers respond to brain stimulation.
* Treatment for focal hand dystonia will not be provided as part of this study.

DETAILED DESCRIPTION:
Objectives:

The purpose of this protocol is to improve understanding of the pathophysiology of dystonia by performing an electrophysiological study using transcranial magnetic stimulation (TMS). The study may reveal new information about the role of gamma frequency oscillations in cortical facilitation in dystonia patients versus healthy volunteer subjects.

The findings of this study may also help to determine if abnormal gamma frequency facilitation might become a potential diagnostic tool for dystonia.

<TAB>

Study population:

1. We intend to study 13 healthy volunteers and 13 patients with a diagnosis of focal hand dystonia. Thirteen subjects for each group are needed based on the power analysis, with an additional three added to the requested accrual to account for drop-outs, yielding a maximum of 16 subjects per group. Up to 15 focal hand dystonia patients and 15 healthy volunteers may be involved in the pilot experiment. The pilot study will be stopped when a trend in the data emerges, so the total number of subjects who participate in the pilot study may end up being less than the maximum requested accrual of 15. Subjects in the pilot experiment are eligible to later participate in the main experiment.

Design:

The subject will be seated with EMG surface electrodes over the First Dorsal Interosseous (FDI) muscle of each hand monitoring muscle activity. The TMS coil will be placed on the surface of the head and the region of motor cortex corresponding to the respective hand muscle control. The baseline motor evoked potential (MEP) for the FDI muscle will be determined by TMS stimulation and EMG monitoring. A pilot experiment will be performed first. Conditioning stimuli, consisting of repetitive subthreshold TMS stimulation with three pulses at one of eight frequencies, will be delivered. A test stimulus, consisting of a single TMS pulse, will follow the conditioning stimuli at the same interval as the conditioning train, but at a suprathreshold intensity in order to determine the MEP amplitude. After every 5 subjects the pilot data will be analyzed to check for a trend in the frequencies that lead to facilitation. Once a trend emerges, the pilot study will be stopped. The four frequencies with the greatest trend toward facilitation will then be selected and used in the main experiment. The main experiment will be performed the same way as the pilot experiment, but will use only the four frequencies found in the pilot experiment. Conditioning stimuli, consisting of repetitive subthreshold TMS stimulation with three pulses at one of the selected four frequencies, will be delivered. A test stimulus, consisting of a single TMS pulse, will follow the conditioning stimuli at the same interval as the conditioning train, but at a suprathreshold intensity in order to determine the MEP amplitude.

Outcome measures:

We will compare the MEP amplitude following TMS conditioning with the baseline MEP amplitude prior to conditioning. The effect on MEP will then be compared between healthy volunteers and dystonia patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Confirmed diagnosis of focal hand dystonia (patients only).
* Between age 18 and 70 years.
* Able to give informed consent
* Right handed
* Agrees to not drink caffeine or alcohol for 48 hours before study session.
* No open scalp wounds or scalp infections.

EXCLUSION CRITERIA:

* Has used illegal drugs within the past 6 months based on history, including but not limited to marijuana, cocaine, methamphetamine, etc. The intent is to exclude those with drug use that may affect study results. Participants who appear to be intoxicated at the time of testing will be rescheduled.
* Has more than 7 alcoholic drinks a week in the case of a woman and 14 alcoholic drinks a week in the case of a man.
* Abnormal findings on neurologic exam (other than dystonia in patient group)
* Has had a brain tumor, a stroke, traumatic brain injury, epilepsy or a history of seizures.
* Has major depression or any major mental disorders (axis I disorders)
* Has a neurologic disorder other than dystonia
* Has had a head injury where there was a loss of consciousness for more than a few seconds.
* Has a pacemaker, intracardiac lines, implanted pumps or stimulators, or has metal objects inside the eye or skull. Dental fillings and dental braces are allowed.
* Has known hearing loss.
* Pregnancy
* Taking any medication that acts as a central nervous system stimulant or that is known to lower seizure threshold, including, imipramine, amitriptyline, doxepine, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, cocaine, (MDMA, ecstasy), phencyclidine (PCP, angel s dust), ketamine, gamma-hydroxybutyrate (GHB), alcohol, theophylline, mianserin, fluoxetine, fluvoxamine, paroxetine, sertraline, citalopram, reboxetine, venlafaxine, duloxetine, bupropion, mirtazapine, fluphenazine, pimozide, haloperidol, olanzapine, quetiapine, aripiprazole, ziprasidone, risperidone, chloroquine, mefloquine, imipenem, penicillin, ampicillin, cephalosporins, metronidazole, isoniazid, levofloxacin, cyclosporin, chlorambucil, vincristine, methotrexate, cytosine arabinoside, BCNU, lithium, anticholinergics, antihistamines, and sympathomimetics.
* Has excessive daytime sleepiness as indicated by a score of 10 or higher on the Epworth Sleepiness Scale.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-02-13; Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Motor evoked potential following TMS conditioning versus the baseline MEP amplitude in dystonia patients and healthy subjects. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Brown P, Farmer SF, Halliday DM, Marsden J, Rosenberg JR. Coherent cortical and muscle discharge in cortical myoclonus. Brain. 1999 Mar;122 ( Pt 3):461-72. doi: 10.1093/brain/122.3.461. PMID 10094255
- [Background] Cardin JA, Carlen M, Meletis K, Knoblich U, Zhang F, Deisseroth K, Tsai LH, Moore CI. Driving fast-spiking cells induces gamma rhythm and controls sensory responses. Nature. 2009 Jun 4;459(7247):663-7. doi: 10.1038/nature08002. Epub 2009 Apr 26. PMID 19396156
- [Background] Crowell AL, Ryapolova-Webb ES, Ostrem JL, Galifianakis NB, Shimamoto S, Lim DA, Starr PA. Oscillations in sensorimotor cortex in movement disorders: an electrocorticography study. Brain. 2012 Feb;135(Pt 2):615-30. doi: 10.1093/brain/awr332. Epub 2012 Jan 16. PMID 22252995